CLINICAL TRIAL: NCT03651440
Title: Effect of PNF and Lumbar Stabilization Exercises on Muscle Strength and Muscle Endurance in Patients With Lumbar Disc Hernia
Brief Title: Effect of PNF and Lumbar Stabilization Exercises on Muscle Strength and Endurance in Lumbar Disc Hernia
Acronym: PNF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Nilay Comuk Balci, associate professor, Baskent University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: KA14/36
Record Dates: First submitted 2018-08-08; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Lumbar Disc Herniation
Keywords: Disc herniation; Endurance; Lumbar stabilization exercise; PNF; Strength
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- lumbar stabilization training (Experimental): lumbar stabilization training exercises
  Interventions: Other: lumbar stabilization training
- PNF training (Experimental): PNF training exercises
  Interventions: Other: PNF
- physical therapy (Experimental): HP,TENS US
  Interventions: Other: Physical Therapy
- control (Sham Comparator): NO APPLİCATİON
  Interventions: Other: Control

INTERVENTIONS:
Other: PNF — PNF
  Arms: PNF training
Other: lumbar stabilization training — lumbar stabilization training
  Arms: lumbar stabilization training
Other: Physical Therapy — Physical Therapy
  Arms: physical therapy
Other: Control — Control group
  Arms: control

SUMMARY:
Background/Objective: This study investigates the effect of lumbar stabilization and proprioceptive neuromuscular facilitation (PNF) training on muscle strength and muscle endurance.

Methods: Sixty-four participants between the ages of 15 and 69 years, graded "protrusion and bulging lumbar herniation" according to the Macnab Classification, were divided into four groups of 16: lumbar stabilization training (strength training, 5 days/week for 4 weeks); PNF training (5 days/week for 4 weeks); physical therapy (hot pack, TENS, ultrasound, 5 days/week for 4 weeks); and control (without any application). Sociodemographic features were recorded and muscle strength tested. Before and after exercise, a visual analog scale (VAS) and Oswestry Disability Index (ODI) were measured by a physical therapist. After 4 weeks, the evaluations were repeated.

Results: There were significant increases in muscle strength and muscle endurance in the lumbar stabilization group, who also showed significant improvement in pain intensity at rest and during activity, and in ODI (p<0.05). Similar results were observed in the PNF group (p<0.05), although not to the same extent. Patients undergoing physical therapy showed significant differences only in pain intensity at rest, at activity, and in ODI (p<0.05).

Conclusion: Undertaking an appropriate physiotherapy and rehabilitation program aiming to reduce waist circumference of patients with low muscle strength and low muscle endurance will help to increase muscle strength and endurance and reduce pain, and contribute toward the correction of functional disabilities.

DETAILED DESCRIPTION:
Lumbar disc herniation (LDH) is a clinical entity characterized by compression of the spinal nerve roots and resultant back and leg pain. Though uncommon, LDH has been reported as a cause of recurrent low back pain.

Although more than 100 risk factors have been identified for LDH, it is difficult to determine a specific etiology. The most important risk factors are intense sporting activity, heavy lifting, frequent rotation of the body, exposure to vibrations, age, tall stature, obesity, smoking, and psychological and genetic factors.

It has been shown that in LDH patients; the strength and endurance of the back and abdominal muscles are reduced, and this aspect has been reported as a major predisposing factor for low back pain. Hence, an exercise program as part of conservative treatment of low back pain and after surgery would be of potential benefit for patients. Twomey and Taylor have shown that behavioral and cognitive principles combined with exercise programs can be effective in reducing disability in patients with chronic low back pain.

The severity of symptoms in disc herniation depends not only on the amount of herniated disc pressure but also on nervous irritability. To reduce the sensitivity of nerve fibers to pain, symptomatic initiatives that include drugs, physical therapy, and psychological methods can be successful. The primary purpose of physical therapy is control of pain and inflammation, and secondarily to improve symptoms such as stiffness in the joints and muscle spasms. Physical therapy also delivers psychological effects. Agents used in physical therapy are generally administered in a combined regimen. We undertook this study to investigate the effect of lumbar stabilization training and proprioceptive neuromuscular facilitation (PNF) training on muscle strength and muscle endurance.

Results The groups showed no difference in demographic and clinical characteristics( p>0.05).

When groups' evaluations before and after treatment were compared, statistically significant differences were found in VAS after treatment (at rest), VAS (at activity), Oswestry Disability Index (ODI), abdominal strength, endurance of back extensor, left hip flexion flexibility, sit and reach flexibility, 60°/sec trunk flexion, 90°/sec trunk extension, 90°/sec trunk flexion, 120°/sec trunk flexion, and 120°/sec trunk extension.

When pairwise comparisons of groups were conducted, there were significant differences in the stabilization group's ODI, left hip flexion flexibility, sit and reach flexibility, 90°/sec trunk extension, and 90°/sec trunk flexion muscle strength values when compared with values in the PNF group.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who were graded as "protrusion and bulging lumbar herniation" according to the Macnab Classification.

Exclusion Criteria:

* Subjects with acute radicular signs or symptoms and those who had radiographic evidence of inflammatory disease affecting the spine, tumor, fracture, spondylolysis, spondylolisthesis, or scoliosis.

Ages: 15 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 64 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2015-01-01 (Actual); Study Completion 2015-01-01 (Actual)

PRIMARY OUTCOMES:
visual analog scale | 4 weeks
  . A standard visual analog scale (VAS) was a used to assess pain. The patients graded their low back pain on a 10-point scale, anchored with the descriptors "no pain" at one end and "pain as bad as it could possibly be" at the other. Maximum pain severity was assessed by a blind-testing physician using the standard VAS

SECONDARY OUTCOMES:
Oswestry Disability Index | 4 weeks
  The Oswestry Disability Questionnare was used to assess pain. The maximum score in this questionnaire is 50, which represents 100% disability.

CONTACTS AND LOCATIONS:
Overall Officials: mitat koz, Prof.Dr., Study Director — Ankara University; nilay comuk balcı, Assoc. Prof, Principal Investigator — Baskent University; nuri çetin, MD.Prof.Dr., Principal Investigator — Baskent University; atakan yılmaz, Pt, Principal Investigator — Baskent University

IPD SHARING:
Plan to Share IPD: Undecided